CLINICAL TRIAL: NCT06228326
Title: KB707-02: A Phase 1/2 Study of Inhaled KB707 in Patients With Advanced Solid Tumor Malignancies Affecting the Lungs
Brief Title: A Study Assessing KB707 for the Treatment of Advanced Solid Tumor Malignancies Affecting the Lungs
Acronym: KYANITE-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB707-02
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer, Non-small Cell; Lung Cancer Metastatic; Solid Tumor, Adult; Advanced Cancer; Lung Cancer (NSCLC)
Keywords: cancer; Krystal Biotech; lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — pembrolizumab; Drug Therapy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohorts 1 through 4 (Experimental): Dose escalation and expansion cohorts: KB707 monotherapy in subjects with solid tumor malignancies affecting the lungs.
  Interventions: Biological: KB707
- Cohort 5 (Experimental): Dose expansion cohort: KB707 administered in combination with Keytruda in approximately 60 subjects with NSCLC.
  Interventions: Biological: KB707; Drug: Pembrolizumab (KEYTRUDA®)
- Cohort 6 (Experimental): Dose expansion cohort: KB707 administered in combination with Keytruda and chemotherapy in approximately 60 subjects with NSCLC.
  Interventions: Biological: KB707; Drug: Pembrolizumab (KEYTRUDA®); Drug: Chemotherapy
- Experimental: Cohort 7 (Experimental): Dose expansion cohort: KB707 administered in combination with docetaxel in approximately 50 subjects with NSCLC.
  Interventions: Biological: KB707; Drug: Docetaxel

INTERVENTIONS:
Biological: KB707 — Genetically modified herpes simplex type 1 virus
Drug: Pembrolizumab (KEYTRUDA®) — PD-1 immune checkpoint inhibitor
  Arms: Cohort 5; Cohort 6
Drug: Chemotherapy — SOC chemotherapy
  Arms: Cohort 6
Drug: Docetaxel — SOC chemotherapy
  Arms: Experimental: Cohort 7

SUMMARY:
The Sponsor is developing KB707, a replication-defective, non-integrating herpes simplex virus type 1 (HSV-1)-derived vector designed to stimulate an anti-tumor immune response through the production of cytokines within the local tumor microenvironment in the lungs. KB707 is administered via nebulization, delivering the therapy directly through the airways to the lungs of subjects with advanced solid tumor malignancies.

This is a Phase 1/2, open-label, multicenter, dose escalation and expansion study designed to evaluate the safety, tolerability, preliminary efficacy, and immunologic effect of KB707.

Monotherapy KB707 dose escalation and expansion cohorts enrolled adults with advanced solid tumor malignancies affecting the lungs who had progressed on standard of care therapy, cannot tolerate standard of care therapy, or refused standard of care therapy. The dose escalation phase (Cohorts 1 and 2) evaluated KB707 monotherapy using a standard 3+3 design, followed by a dose expansion phase (Cohort 4) to further evaluate the selected dose. Subjects received inhaled KB707 weekly for three weeks, then every three weeks. The dose escalation portion of the study is now complete, and the selected dose is being evaluated in the expansion phase.

Combination regimens with a selected (fixed) dose of KB707 are being evaluated in subjects with advanced or metastatic non-small cell lung cancer (NSCLC). Subjects in Cohorts 5 and 6 are receiving inhaled KB707 once every 2 weeks (q2w), delivered in combination with Keytruda once every 6 weeks. Subjects in Cohort 7 are receiving inhaled KB707 in combination with docetaxel once every 3 weeks.

All subjects will be treated until tumor progression, death, unacceptable toxicity, symptomatic deterioration, achievement of maximal response, subject choice, Investigator decision to discontinue treatment, or the Sponsor determines to terminate the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 years or older at the time of informed consent
* Life expectancy >12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have at least one measurable lung lesion per RECIST v1.1 at Screening
* Cohorts 1 through 4 only: Histologically confirmed diagnosis of advanced solid tumor malignancy affecting the lungs and the individual has progressed on standard of care therapy, cannot tolerate standard of care therapy, refused standard of care therapy, or has no standard of care therapy.
* Cohorts 5, 6, and 7 only: (1) Histologically or cytologically confirmed diagnosis of stage 3 or 4 NSCLC, as per American Joint Committee on Cancer (AJCC) staging system (8th edition) and (2) Subject must meet the following criteria of prior lines of therapy:

  1. Subject has previously received no more than one line of prior immune checkpoint inhibitor (ICI) with or without platinum-based chemotherapy, or no more than two prior lines of therapy when given the ICI and platinum-based chemotherapy sequentially as two separate lines.
  2. Subjects with an actionable mutation (e.g., EGFR, KRAS, ALK, or ROS1 genomic alteration), are permitted to have received one additional line of approved targeted therapy.

Key Exclusion Criteria:

* Not fully recovered from prior surgery or radiotherapy, including all radiation-related toxicities
* The subject is pregnant, nursing, or plans to become pregnant during study treatment and through three months after the last dose of KB707
* Have known history of positive human immunodeficiency virus (HIV 1/2)
* Cohorts 5, 6, and 7 only:

  1. Subject has a known additional malignancy that is progressing or requires active treatment
  2. Subject has active brain metastases or leptomeningeal metastases
  3. Prior anti-PD-1/PD-L1 therapy was intolerable and required discontinuation of treatment
  4. Subject has active, known, or suspected autoimmune disease requiring systemic treatment
  5. Subject has known acute or chronic hepatitis
  6. Subject has active pneumonitis or history of ICI-induced pneumonitis that required steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of inhaled KB707 based upon assessment of adverse events (AE) | up to 36 months
  Percentage of subjects with treatment-related AEs as assessed by NCI-CTCAE v5

SECONDARY OUTCOMES:
To evaluate whether the proposed dose ranges include the maximum tolerated dose of KB707 as determined by incidence of dose limiting toxicities (DLTs) | up to 36 months
  Incidence of dose limiting toxicity (DLT) by dose cohorts
To evaluate the preliminary efficacy of inhaled KB707 as determined by overall response rate (ORR) | up to 36 months
  Percentage of ORR for all participants

CONTACTS AND LOCATIONS:
Overall Officials: David Chien, MD, Study Director — Senior Vice President of Clinical Development
Locations (14):
- United States (14):
  - XCancer Research Network/Dothan Hematology & Oncology, Dothan, Alabama
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Precision NextGen Oncology, Beverly Hills, California
  - Emad Ibrahim MD Inc, Redlands, California
  - BRCR Global, Weston, Florida
  - IU Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - Ochsner/MD Anderson Cancer Center, New Orleans, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - Gabrail Cancer Center Research, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nasville, Tennessee
  - Renovatio Clinical, El Paso, Texas
  - Renovatio Clinical, The Woodlands, Texas